CLINICAL TRIAL: NCT00214461
Title: A Phase I Randomized, Placebo-Controlled, Double-Blind, Dose Ranging Study of the Safety, Tolerability and Immunogenicity of a Clostridium Difficile Toxoid Vaccine, Alum Adsorbed, in Healthy Elderly Volunteers (> or =65 Years)
Brief Title: Safety, Tolerability, and Immunogenicity of a Clostridium Difficile Toxoid Vaccine in Healthy Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-030-009
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Clostridium Infections
Keywords: Clostridium difficile
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Vaccine Group (Placebo Comparator): Participants will receive a dose of vaccine diluent (placebo) on Days 0, 28 and 56, respectively.
  Interventions: Biological: Vaccine diluent buffer (Placebo)
- Low Dose Vaccine Group (Experimental): Participants will receive a dose of vaccine containing of 2 µg Clostridium Difficile toxoid on Days 0, 28 and 56, respectively.
  Interventions: Biological: C. difficile toxoid vaccine (2 µg)
- Medium dose vaccine group (Experimental): Participants will receive a dose of vaccine containing of 10 µg Clostridium Difficile toxoid on Days 0, 28 and 56, respectively.
  Interventions: Biological: C. difficile toxoid vaccine (10 µg)
- High dose vaccine group (Experimental): Participants will receive a dose of vaccine containing of 50 µg Clostridium Difficile toxoid on Days 0, 28 and 56, respectively.
  Interventions: Biological: C. difficile toxoid vaccine (50 µg)

INTERVENTIONS:
Biological: Vaccine diluent buffer (Placebo) — 0.5 mL, Intramuscular on Day 0, Day 28, and Day 56, respectively.
  Arms: Placebo Vaccine Group
Biological: C. difficile toxoid vaccine (2 µg) — 0.5 mL, Intramuscular on Day 0, Day 28, and Day 56, respectively.
  Arms: Low Dose Vaccine Group
Biological: C. difficile toxoid vaccine (10 µg) — 0.5 mL, Intramuscular on Day 0, Day 28 and Day 56, respectively.
  Arms: Medium dose vaccine group
Biological: C. difficile toxoid vaccine (50 µg) — 0.5 mL, Intramuscular on Day 0, Day 28, and Day 56, respectively.
  Arms: High dose vaccine group

SUMMARY:
The purpose of this study is to determine the safety and tolerability of a modified C. difficile vaccine at 3 dose levels compared with a placebo control administered via intramuscular injection in healthy elderly subjects aged > or = 65 years. This is the companion study to H-030-008, in which healthy younger adults have already been dosed.

DETAILED DESCRIPTION:
Clostridium difficile is the leading infectious cause of nosocomial diarrhea in developed countries. Hospital outbreaks of Clostridium difficile-associated diarrhea (CDAD) are associated with substantial patient morbidity and mortality. Conventional therapy with antibiotics often results in secondary infection with resistant organisms or clinical relapse after discontinuation of the antimicrobial course. New strategies are needed to limit the impact of this opportunistic pathogen. Considerable evidence exists that immunity against C. difficile toxins may be effective in controlling CDAD. 48 subjects will be enrolled to receive one of three dose levels of modified C difficile vaccine or placebo administered on a 3-dose schedule. The study consists of a 30-day screening period, a 70-day treatment period, one follow-up phone interview 2 months after the last vaccination, and one follow-up clinic visit 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females, > or = 65 years
* In good general health
* Clinical lab tests within normal range
* Females must be post-menopausal
* Able and willing to participate for duration of study and must not participate in any other experimental study for at least 60 days after receiving the last dose of study vaccine

Exclusion Criteria:

* Evidence of C. difficile infection
* Evidence of any previous antibiotic-associated diarrhea
* Active or inactive inflammatory bowel disease, irritable colon syndrome, chronic abdominal pain or other chronic diarrhea
* History of malignancy within 5 years
* History of anaphylaxis, asthma or severe vaccine or severe allergic drug reaction
* Known or suspected history of immunodeficiency
* Active or inactive immune-mediated or inflammatory disease
* History of drug or alcohol abuse disorders;
* Serology positive for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Receipt of antibiotic therapy or an investigational drug within prior 30 days
* Blood or organ donation within prior 30 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Richard Greenberg, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - University of Kentucky, Lexington, Kentucky

REFERENCES:
- [Derived] Greenberg RN, Marbury TC, Foglia G, Warny M. Phase I dose finding studies of an adjuvanted Clostridium difficile toxoid vaccine. Vaccine. 2012 Mar 16;30(13):2245-9. doi: 10.1016/j.vaccine.2012.01.065. Epub 2012 Feb 2. PMID 22306375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 01 November 2005 to 11 October 2006 in 3 medical centers in the US.
Pre-assignment Details: A total of 48 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Placebo Vaccine Group: Participants who received a dose of placebo, on Days 0, 28, and 56, respectively.
- Low-dose C. Difficile Vaccine Group: Participants who received a dose of vaccine containing 2 µg C. difficile toxoid on Days 0, 28, and 56, respectively.
- Medium-dose C. Difficile Vaccine Group: Participants who received a dose of vaccine containing 10 µg C. difficile toxoid on Days 0, 28, and 56, respectively.
- High-dose C. Difficile Vaccine Group: Participants who received a dose of vaccine containing 50 µg, C. difficile vaccine on Days 0, 28, and 56, respectively.
Period: Overall Study
Arm/Group | Placebo Vaccine Group | Low-dose C. Difficile Vaccine Group | Medium-dose C. Difficile Vaccine Group | High-dose C. Difficile Vaccine Group
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 10 | 11
Not Completed | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Vaccine Group | Low-dose C. Difficile Vaccine Group | Medium-dose C. Difficile Vaccine Group | High-dose C. Difficile Vaccine Group | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 12 | 12 | 12 | 12 | 48
Age Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (3.59) | 72.2 (5.32) | 75.5 (6.47) | 68.9 (4.32) | 71.4 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 7 | 26
  Male | 6 | 4 | 7 | 5 | 22
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 48

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Achieving Seroconversion of Serum Immunoglobulin G (IgG) After Vaccination With Either a Formulation of C. Difficile Toxoid Vaccine or a Placebo Vaccine.
Description: Seroconversion was defined as a ≥ 4-fold increase from baseline in a subject's specific IgG levels: Serum Levels of Anti-toxin Immunoglobulin (IgG) against toxin A and toxin B in enzyme units (EU) were assessed by enzyme linked immunosorbent assay (ELISA).
Time Frame: Day up to Day 236 post first vaccination
Population: Serum anti-toxin levels were assessed in the fully evaluable (Per-Protocol) population.
Measure: Number; unit: Participants
Arm/Group | Placebo Vaccine Group | Low-dose C. Difficile Vaccine Group | Medium-dose C. Difficile Vaccine Group | High-dose C. Difficile Vaccine Group
Number analyzed (Participants) | 11 | 12 | 9 | 11
Participants
  Toxin A: Day 14 | 0 | 0 | 1 | 3
  Toxin A: Day 28 | 0 | 2 | 2 | 4
  Toxin A: Day 56 | 0 | 6 | 8 | 11
  Toxin A: Day 70 | 0 | 11 | 9 | 11
  Toxin A: Day 236 | 0 | 3 | 4 | 5
  Toxin B: Day 14 | 0 | 2 | 2 | 4
  Toxin B: Day 28 | 0 | 3 | 2 | 5
  Toxin B: Day 56 | 0 | 4 | 4 | 5
  Toxin B: Day 70 | 0 | 7 | 5 | 8
  Toxin B: Day 236 | 0 | 3 | 1 | 3

2. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events Post-vaccination With Either One of Three Formulations of the Clostridium Difficile Vaccine or a Placebo Vaccine.
Time Frame: Day 0 to up to 70 days post first vaccination
Population: Safety assessments were on the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo Vaccine Group | Low-dose C. Difficile Vaccine Group | Medium-dose C. Difficile Vaccine Group | High-dose C. Difficile Vaccine Group
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Injection site pain | 3 | 8 | 4 | 8
  Eosinophil count increased | 4 | 5 | 3 | 5
  White blood cells urine positive | 3 | 1 | 5 | 6
  Fatigue | 2 | 3 | 2 | 4
  Myalgia | 2 | 4 | 1 | 4
  Arthralgia | 2 | 5 | 1 | 1
  Injection site erythema | 1 | 3 | 1 | 3
  Headache | 2 | 3 | 2 | 1
  Back pain | 1 | 3 | 0 | 2
  Blood urea increased | 1 | 0 | 3 | 2
  Diarrhoea | 1 | 2 | 2 | 1
  White blood cell count increased | 2 | 0 | 2 | 2
  Protein urine present | 0 | 0 | 3 | 2
  Vomiting | 1 | 2 | 1 | 1
  Anorexia | 2 | 1 | 0 | 2
  Red blood cells urine positive | 2 | 0 | 1 | 2
  Nasopharyngitis | 0 | 1 | 2 | 1
  Blood bilirubin increased | 0 | 0 | 2 | 1
  Blood potassium increased | 0 | 0 | 1 | 2
  Haemoglobin decreased | 0 | 1 | 2 | 0
  Injection site warmth | 0 | 2 | 0 | 1
  Red blood cell count decreased | 2 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of vaccination (Day 0) for up to 1 year post-vaccination
Arm/Group | Placebo Vaccine Group | Low-dose C. Difficile Vaccine Group | Medium-dose C. Difficile Vaccine Group | High-dose C. Difficile Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 2/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 12/12 | 11/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Vaccine Group (N=12) | Low-dose C. Difficile Vaccine Group (N=12) | Medium-dose C. Difficile Vaccine Group (N=12) | High-dose C. Difficile Vaccine Group (N=12)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo Vaccine Group (N=12) | Low-dose C. Difficile Vaccine Group (N=12) | Medium-dose C. Difficile Vaccine Group (N=12) | High-dose C. Difficile Vaccine Group (N=12)
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 2 | 4
Induration (General disorders) | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 3 | 1 | 3
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 1 | 0 | 1
Injection site nodule (General disorders) | 0 | 1 | 0 | 0
Injection site oedema (General disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 3 | 8 | 4 | 8
Injection site pruritus (General disorders) | 0 | 1 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 1
Injection site swelling (General disorders) | 0 | 1 | 0 | 1
Injection site warmth (General disorders) | 0 | 2 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 1 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1 | 2
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 3 | 2
Electrocardiogram ST T Change (Investigations) | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 4 | 5 | 3 | 5
Glucose urine (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 2 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 1
Prostate examination abnormal (Investigations) | 0/6 | 0/4 | 0/7 | 1/5
Protein urine present (Investigations) | 0 | 0 | 3 | 2
Red blood cell count decreased (Investigations) | 2 | 0 | 1 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 2 | 0 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 2 | 0 | 2 | 2
White blood cells urine positive (Investigations) | 3 | 1 | 5 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 2 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0/6 | 0/4 | 1/7 | 0/5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolarygeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications